CLINICAL TRIAL: NCT00017914
Title: Studies in the Natural History and Pathogenesis of Childhood-Onset and Adult-Onset Idiopathic Inflammatory Myopathies
Brief Title: Adult and Juvenile Myositis
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940165; 94-E-0165; NCT00001374 (obsolete NCT alias)
Record Dates: First submitted 2001-06-19; First posted 2001-06-20 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-06-27

CONDITIONS: Dermatomyositis; Polymyositis; Inclusion Body Myositis
Keywords: Adult and Pediatric Disease; Autoimmunity Pathogenesis; Disease Assessment; Genetic and Environmental Risk Factors; Myositis; Natural History
MeSH Terms: conditions — Dermatomyositis; Polymyositis; Myositis, Inclusion Body; Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteer: Healthy subject who has not received anti-inflammatory medications and should not has undergone surgery or any major trauma within the 8 weeks prior to enrollment.
- Myositis Patient: Patient should have documented evidence that he/she meets criteria for an idiopathic inflammatory myopathy (IIM)
- Non-Myositis Patient: Patients with other myopathies/autoimmune diseases/complications similar to myositis patients. Close relatives of IIM patients (affected or unaffected siblings, children, parents, grandparents)

SUMMARY:
This study will evaluate subjects with adult- and childhood-onset myositis to learn more about their cause and the immune system changes and medical problems associated with them. Myositis is an inflammatory muscle disease that can damage muscles and other organs, resulting in significant disability.

Children or adults with polymyositis or dermatomyositis or a related condition may be evaluated under this study. Healthy children or adults will also be enrolled as "controls," for comparison of test results.

All patients will undergo a complete history (including completing some questionnaires) and physical examination, review of medical records, and blood and urine tests. Patients may then choose to participate in an additional 1- to 5-day evaluation, which will include some or all of the following diagnostic, treatment or research procedures:

1. Standardized muscle strength testing, range of motion of joints and walking (gait) analysis by a physiotherapist; completion of a questionnaire regarding ability to perform daily tasks
2. Skin assessment, possibly including photographs of lesions and a skin biopsy (removal of a small skin sample under local anesthetic)
3. Magnetic resonance imaging (scans that use magnetic fields to visualize tissues) of leg muscles
4. Swallowing studies, including a physical examination and questionnaire on swallowing ability, studies of tongue strength, and ultrasound imaging during swallowing, and possibly, a modified barium swallow
5. Voice and speech assessment, possibly including computerized voice analysis and laryngoscopy-analysis of the larynx (voice box) using a small rigid scope with a camera placed in the mouth to view and record vocal cord function
6. Pulmonary function tests (measurement of air moved into and out of the lungs, using a breathing machine) to evaluate lung function and, possibly, chest X-ray
7. Electrocardiogram (measurement of the electrical activity of the heart) and, possibly, echocardiogram (ultrasound imaging of the heart)
8. Endocrine evaluation
9. Eye examination, in patients with vision loss or other eye symptoms
10. Nutrition assessment to evaluate muscle mass and muscle wasting, including tape measurements or bioelectric impedance testing, a painless procedure in which wires are attached to the extremities with a sticky paste.
11. Muscle ultrasound.
12. Electromyography (record of the electrical activity of muscles)
13. Muscle or skin biopsy (removal of a small piece of muscle tissue for microscopic examination)

All patients may have only a one-time evaluation or may return for one follow-up evaluations (either the 1-day or 3- to 5-day evaluation) over a 1-year period.

Healthy children will undergo a medical history and brief physical examination; blood and urine tests; speech and swallowing studies including questionnaires and physical examination, tongue strength, and ultrasound study; and bioelectric impedance testing. Children 8 to 18 years old may also have exercise testing.

DETAILED DESCRIPTION:
This study will evaluate subjects with adult- and childhood-onset myositis to learn more about their cause and the immune system changes and medical problems associated with them. Myositis is an inflammatory muscle disease that can damage muscles and other organs, resulting in significant disability.

Children or adults with polymyositis or dermatomyositis or a related condition may be evaluated under this study. Healthy children or adults will also be enrolled as "controls," for comparison of test results.

All patients will undergo a complete history (including completing some questionnaires) and physical examination, review of medical records, and blood and urine tests. Patients may then choose to participate in an additional 1- to 5-day evaluation, which will include some or all of the following diagnostic, treatment or research procedures:

1. Standardized muscle strength testing, range of motion of joints and walking (gait) analysis by a physiotherapist; completion of a questionnaire regarding ability to perform daily tasks
2. Skin assessment, possibly including photographs of lesions and a skin biopsy (removal of a small skin sample under local anesthetic)
3. Magnetic resonance imaging (scans that use magnetic fields to visualize tissues) of leg muscles
4. Swallowing studies, including a physical examination and questionnaire on swallowing ability, studies of tongue strength, and ultrasound imaging during swallowing, and possibly, a modified barium swallow
5. Voice and speech assessment, possibly including computerized voice analysis and laryngoscopy-analysis of the larynx (voice box) using a small rigid scope with a camera placed in the mouth to view and record vocal cord function
6. Pulmonary function tests (measurement of air moved into and out of the lungs, using a breathing machine) to evaluate lung function and, possibly, chest X-ray
7. Electrocardiogram (measurement of the electrical activity of the heart) and, possibly, echocardiogram (ultrasound imaging of the heart)
8. Endocrine evaluation
9. Eye examination, in patients with vision loss or other eye symptoms
10. Nutrition assessment to evaluate muscle mass and muscle wasting, including tape measurements or bioelectric impedance testing, a painless procedure in which wires are attached to the extremities with a sticky paste.
11. Muscle ultrasound.
12. Electromyography (record of the electrical activity of muscles)
13. Muscle or skin biopsy (removal of a small piece of muscle tissue for microscopic examination)

All patients may have only a one-time evaluation or may return for one follow-up evaluations (either the 1-day or 3- to 5-day evaluation) over a 1-year period.

Healthy children will undergo a medical history and brief physical examination; blood and urine tests; speech and swallowing studies including questionnaires and physical examination, tongue strength, and ultrasound study; and bioelectric impedance testing. Children 8 to 18 years old may also have exercise testing.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Patients with Myositis:

Inclusion Criteria:

All patients should have age range 2-100 years.

All Patients admitted to the study must satisfy at least one of the following criteria among item 1 (A or B or C) OR item 2 (A or B or C) AND item 3:

1. Patient has documented evidence that he/she meets criteria for an idiopathic inflammatory myopathy

   A. Possible, probable or definite adult or juvenile polymyositis or dermatomyositis by Bohan and Peter criteria

   B. Possible, probable or definite inclusion body myositis by Griggs and/or ENMC criteria

   C. Has an idiopathic inflammatory myopathy that does not meet these criteria, including common or rarer forms of myositis such as cancer- associated, focal, orbital, eosinophilic myositis, macrophagic, proliferative, etc.
2. Has one of the following conditions:

2A. Have a disorder that is related to an idiopathic inflammatory myopathy, that may include:

* Inflammatory and non-inflammatory myopathies:
* Mimicking and related skin disorders:
* Disorders of the complications of myositis (including interstitial lung disease, calcifying disorders, cardiomyopathies, etc.):
* Overlapping autoimmune diseases that may be associated with myositis
* Patients with muscle and/or skin inflammation and documented environmental exposures:
* Patients with myositis or complications of myositis and suspected genetic disorders:
* Patients with undifferentiated connective tissue disease
* Patients with signs or symptoms of myositis (such as weakness, skin rashes, interstitial lung disease) or laboratory abnormalities (such as elevated CK or muscle biopsy with myopathic features) who do not have an established diagnosis of myositis for them to be evaluated to establish a diagnosis

  3. Ability of patient or parent/guardian to give informed consent to all or part of the study after full information has been provided.

Exclusion Criteria:

1. Patients <2 years or >100 years will be excluded.
2. Any conditions in which the drawing of the amount of blood required or undergoing procedures needed for the study is not deemed medically appropriate by the treating physician or the principal investigator.

For females of childbearing potential who are pregnant, they will be permitted to enroll, but would be excluded from radiographic procedures involving radiation or greater than minimal risk procedures, including obtaining biopsies.

Relatives of Patients with Myositis:

For patients with at least one first-degree relative affected with IIIM, all available first-degree relatives (affected and unaffected) are eligible to participate in the genetics portion of the protocol. For patients in which two or more first degree relatives are affected with myositis, any available close relatives (affected or unaffected parents, siblings or children, as well as grandparents and grandchildren, or other close relatives, when available) are eligible to participate in the genetics portion of the protocol.

Inclusion criteria:

1. First or more distant relative of a proband with myositis, for genetics studies.
2. Ability of patient or parent/guardian to give informed consent to all or part of the study after full information has been provided.

Exclusion Criteria:

1. Patients <2 years or >100 years will be excluded.
2. Any conditions in which the drawing of the amount of blood required or undergoing procedures needed for the study is not deemed medically appropriate by the treating physician or the principal investigator.
3. Pregnancy (females of childbearing potential). Verbal confirmation they are not pregnant.

Healthy Volunteers:

Inclusion Criteria:

1. Healthy volunteer subjects for biomarker studies will be gender and age-matched (within 5 years) with a myositis patient, as reasonably close as possible.
2. Volunteer is not related to a myositis patient who is enrolled in the study
3. Volunteer is in good health, without a recognized systemic rheumatic disorder, autoimmune disease, immune medicated disease, or cancer, and is not taking any anti-inflammatory medicines, including nonsteroidal anti-inflammatory drugs (NSAIDS) or corticosteroids
4. Volunteer or volunteer s parent/guardian could give assent/informed consent to all or part of the study after full information has been provided

Exclusion Criteria:

If Any "Yes" answer patient is not eligible for study

1. Volunteer has undergone surgery or had a major trauma within the past 2 months
2. Volunteer used anti-inflammatory medications within the past 8 weeks of enrollment, including not currently receiving nonsteroidal anti-inflammatory drugs or corticosteroids
3. Volunteer has been diagnosed with a chronic infectious illness, inflammatory disease, malignancy, cardiac or pulmonary disease, muscle disorder, clotting disorder, metabolic disorder, systemic rheumatic or autoimmune disease, or immune-mediated disease
4. Volunteer is pregnant (verbally screened for females of childbearing potential)
5. Volunteer has a medical illness that in the judgement of the investigators does not allow safe blood draws or other clinical evaluations needed for study participation
6. Volunteer is cognitively impaired
7. Volunteer and or the volunteer's parents/legal guardian is unable or unwilling to give informed consent/assent
8. Volunteer has functional limitations
9. Volunteer has joint or muscle problems

Note that the following screening activities may be performed to determine subject eligibility:

* Email, written, or telephone communications with prospective subjects
* Review of existing medical records
* Review of existing imaging studies
* Review of existing photographs or videos
* Review of existing pathology specimens/reports from a specimen obtained for diagnostic purposes

If a participant is ineligible and willing, their contact information- including name, phone numbers, emails, best times to reach, and potential diagnosis- may be shared with other NIH investigators if the participant may be eligible to participate in those studies.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1- Any patient who has documented evidence that he/she meets criteria for an idiopathic inflammatory myopathy; 2- Any patient who has been diagnosed with inflammatory/non-inflammatory myopathies, mimicking and related skin disorders, disorders of complications of myositis, overlapping autoimmune diseases that may be associated with myositis, patients with muscle and/or skin inflammation and documented environmental exposures, patients with myositis or complications of myositis and suspected genetic disorders, patients with undifferentiated connective tissue disease, patients with signs or symptoms of myositis or laboratory abnormalities who do not have an established diagnosis of myositis for them to be evaluated to establish a diagnosis; 3- Close relatives of patients with at least one first-degree relative affected with IIIM (affected or unaffected siblings, children, parents, grandparents) can participate in the genetics portion of the protocol; 4- Healthy control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 1995-06-07 (Actual)

PRIMARY OUTCOMES:
Physician Global Assessment Form | At enrollment and each study visit
  1- A secure internet accessible IMACS Outcomes Data Repository of core set disease activity, damage and quality of life measures has been established for adult and juvenile myositis patients as part of IMACS. 2- Compare the clinical and immunopathogenic features of childhood and adult IIM to determine the differences of IIM in these two populations referred to NIH 3- investigate the immunopathogenesis and immunogenetics of IIM.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa G Rider, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina
  - Texas Scottish Rite Hospital, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller FW, Lamb JA, Schmidt J, Nagaraju K. Risk factors and disease mechanisms in myositis. Nat Rev Rheumatol. 2018 Apr 20;14(5):255-268. doi: 10.1038/nrrheum.2018.48. PMID 29674613
- [Background] Miller FW, Chen W, O'Hanlon TP, Cooper RG, Vencovsky J, Rider LG, Danko K, Wedderburn LR, Lundberg IE, Pachman LM, Reed AM, Ytterberg SR, Padyukov L, Selva-O'Callaghan A, Radstake TR, Isenberg DA, Chinoy H, Ollier WE, Scheet P, Peng B, Lee A, Byun J, Lamb JA, Gregersen PK, Amos CI; Myositis Genetics Consortium. Genome-wide association study identifies HLA 8.1 ancestral haplotype alleles as major genetic risk factors for myositis phenotypes. Genes Immun. 2015 Oct;16(7):470-80. doi: 10.1038/gene.2015.28. Epub 2015 Aug 20. PMID 26291516
- [Background] Rider LG, Aggarwal R, Machado PM, Hogrel JY, Reed AM, Christopher-Stine L, Ruperto N. Update on outcome assessment in myositis. Nat Rev Rheumatol. 2018 May;14(5):303-318. doi: 10.1038/nrrheum.2018.33. Epub 2018 Apr 12. PMID 29651119
- [Background] Sparling AC, Ward JM, Sarkar K, Schiffenbauer A, Farhadi PN, Smith MA, Rahman S, Zerrouki K, Miller FW, Li JL, Casey KA, Rider LG. Neutrophil and mononuclear leukocyte pathways and upstream regulators revealed by serum proteomics of adult and juvenile dermatomyositis. Arthritis Res Ther. 2024 Nov 11;26(1):196. doi: 10.1186/s13075-024-03421-7. PMID 39529136
- [Background] Burbelo PD, Huapaya JA, Khavandgar Z, Beach M, Pinal-Fernandez I, Mammen AL, Chiorini JA, Noroozi Farhadi P, Miller FW, Schiffenbauer A, Sarkar K, Warner BM, Rider LG. Quantification of autoantibodies using a luminescent profiling method in autoimmune interstitial lung disease. Front Immunol. 2024 Oct 25;15:1462242. doi: 10.3389/fimmu.2024.1462242. eCollection 2024. PMID 39524452
- [Background] Sherman MA, Noroozi Farhadi P, Pak K, Trieu EP, Sarkar K, Targoff IN, Neely ML, Mammen AL, Rider LG; Childhood Myositis Heterogeneity Collaborative Study Group. Myositis-Associated Autoantibodies in Patients With Juvenile Myositis Are Associated With Refractory Disease and Mortality. Arthritis Rheumatol. 2024 Jun;76(6):963-972. doi: 10.1002/art.42813. Epub 2024 Mar 12. PMID 38272842
- [Background] Ward JM, Ambatipudi M, O'Hanlon TP, Smith MA, de Los Reyes M, Schiffenbauer A, Rahman S, Zerrouki K, Miller FW, Sanjuan MA, Li JL, Casey KA, Rider LG. Shared and Distinctive Transcriptomic and Proteomic Pathways in Adult and Juvenile Dermatomyositis. Arthritis Rheumatol. 2023 Nov;75(11):2014-2026. doi: 10.1002/art.42615. Epub 2023 Aug 13. PMID 37229703
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1994-E-0165.html